CLINICAL TRIAL: NCT01929525
Title: Effectiveness of Silver Nitrate Solution in the Treatment of Anal Fistula: A Novel Strategy for Managing Anal Fistula
Brief Title: Effectiveness of Silver Nitrate Solution in the Treatment of Anal Fistula
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, M.Umit UGURLU, Assistant profesor of surgery, Marmara University
Other Study IDs: MarmaraUSM
Record Dates: First submitted 2013-08-19; First posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Silver Nitrate: Irrigation of fistula tract with 1% silver nitrate solution for all patients who accepts the study and signed the written informed consent form.

SUMMARY:
Effectiveness of silver nitrate solution in treatment of anal fistula is is aimed to be investigated.

DETAILED DESCRIPTION:
The anal fistula is a granulation tissue-lined tract, we thought of a way to ablate this granulation tissue using a chemical agent, which would eventually induce healing with fibrosis and closure of the tract without any surgical intervention. Aiming to reduce the surgery related complications; we investigated the effectiveness of silver nitrate solution as a chemical agent in the treatment of anal fistula.

ELIGIBILITY:
Inclusion Criteria:

All patients with the diagnosis of anal fistula Patients with recurrence

Exclusion Criteria:

Patients who do not sign the informed consent

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of anal fistula
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Number of anal fistula patients treated with silver nitrate solution. | 1 year
  The primary end point in the study was to assess the efficacy of the silver nitrate in the treatment of anal fistula. The number of anal fistula patients who are treated with silver nitrate solution will be calculated. The role of silver nitrate solution in anal fistula treatment will be investigated

SECONDARY OUTCOMES:
Therapeutic factors | 1 year
  The secondary end point was to identify the clinical and therapeutic factors that significantly affect the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: S.CUMHUR YEGEN, MD, Study Chair — Marmara University
Locations (1):
- MarmaraUSM, Istanbul, Istanbul, Turkey (Türkiye)